CLINICAL TRIAL: NCT05194332
Title: Transcranial Low Intensity Focused Ultrasound Neuromodulation as a Probe to Study Human Emotion and Cognitive Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jair Soares, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-21-0570
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Depressive Disorder, Major
Keywords: depression; mental illness
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- LIFUP sonication to the amygdala (Experimental)
  Interventions: Device: LIFUP sonication to the amygdala

INTERVENTIONS:
Device: LIFUP sonication to the amygdala — LIFUP sonication to amygdala will be performed.

SUMMARY:
The purpose of this study is to assess the low-intensity focused ultrasound pulsation (LIFUP) neuromodulation on emotion processing in healthy individuals, and to assess the overall safety of the LIFUP to stimulate or inhibit brain activity in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Must be right-handed
* Must be illicit drug-free at the time of scanning as appropriate (verified by negative urine drug screen)
* Must be healthy (without medical, neurological, psychiatric illness)
* Must be psychotropic medication free (≥ 14 days)

Exclusion Criteria:

* Must not be a smoker
* Females must not be pregnant or nursing
* Must not suffer from claustrophobia
* Must not meet exclusion criteria for MRI scanning (i.e., non-fixed magnetizable objects)
* Must not have ongoing, chronic, or relapsing/remitting medical, psychiatric,or neurological illness as determined by a combination of history, medical record, and/or examination.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in amygdala activity indicated by functional magnetic resonance imaging (fMRI) scan blood oxygen-level-dependent (BOLD) signal | baseline, 5 mins post-LIFUP sonication
Changes in brain resting state functional network as indicated by fMRI scan connectivity measures | baseline, 10-20 mins post-LIFUP sonication

SECONDARY OUTCOMES:
Change in performance on Reward Task | baseline, 1-hour post-LIFUP sonication
Tolerability of LIFUP sonication as assessed number of adverse events | baseline, immediately after LIFUP sonication

CONTACTS AND LOCATIONS:
Overall Officials: Jair Soares, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No